CLINICAL TRIAL: NCT05100095
Title: Hypofractionated Radiation Therapy for Merkel Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0789; NCI-2021-12100 (Other: NCI-Clinical Trials Reporting)
Record Dates: First submitted 2021-10-15; First posted 2021-10-29 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Radiation therapy (Experimental): Patients receive radiation therapy in 10 daily fractions (M-F) over 2 weeks.
  Interventions: Drug: Radiation therapy

INTERVENTIONS:
Drug: Radiation therapy — Hypofractionated radiation therapy to the primary tumor and/or lymph nodes

SUMMARY:
This phase II trial tests whether hypofractionated radiation works to treat patients with Merkel cell carcinoma. Radiation therapy uses high energy radio waves to kill cancer cells and shrink tumors. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may be more convenient for patients and less immunosuppressive.

DETAILED DESCRIPTION:
* To estimate the 2-year local control rate for adjuvant hypofractionated RT to the primary tumor bed.
* To estimate the 2-year nodal control rate for adjuvant hypofractionated RT to the primary draining nodal basin.

Secondary Objectives

* To determine MCC disease outcomes including:time to non-nodal locoregional recurrence, time to nodal recurrence, time to distant mestasis, disease-free-survival and disease-specific survival for patients receiving hypofractionated adjuvant RT.
* To assess acute and late RT associated toxicity within or neighboring the radiated field.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed MCC.
* Patients must have no evidence of distant metastasis as determined by clinical examination and any form of imaging.
* If planned for adjuvant primary tumor radiation therapy a patient should have had surgical excision of a primary MCC tumor within 4 months of starting RT.
* If planned for adjuvant nodal radiation therapy a patient should have had:

  * Prior positive sentinel lymph node biopsy with any degree of nodal involvement within 4 months of starting RT and no completion nodal dissection, or
  * Lymph node dissection within 4 months of starting RT and high risk nodal disease (receipt of neoadjuvant immunotherapy, ECE, >1 involved node, >1 cm nodal disease).
* Immunotherapy is permitted at any time and may specifically be administered prior to RT, concurrent with RT or after RT.
* Age ≥18 years because MCC is extremely rare in patients <18 years of age and RT is considered high risk in this population due to risk of secondary malignancy and potentially growing tissues that may be adversely impacted by RT.
* ECOG performance status ≤3.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* RT is a known teratogen. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (refer to MDA Policy CLN 1114) This includes all female patients, between the onset of menses and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following: • Postmenopausal (no menses in greater than or equal to 12 consecutive months). • History of hysterectomy or bilateral salpingo-oophorectomy. • Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy). • History of bilateral tubal ligation or another surgical sterilization procedure. Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of RT.
* Ability to understand and the willingness to sign a written informed consent document.

Expansion cohort

• Patient would have received <50.4 Gy using conventional radiotherapy dose-fractionation if not enrolled.

Exclusion Criteria:

* Previous radiation therapy to the site of planned primary or nodal radiation treatment such that the prior site of treatment would be encompassed by the radiation field needed to treat the current cancer. In other words, treatment on this trial would require re-irradiation of tissues.
* Patients with distant metastases
* Pregnant women are excluded from this study because RT is a known teratogen.
* Patients who are less than 18 years of age becase RT is extremely rare in this population and the treatment agent is a known carcinogen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
To establish the 2-year local control rate for adjuvant hypofractionated RT to the primary tumor bed. And to establish the 2-year nodal control rate for adjuvant hypofractionated RT to the primary draining nodal bed. | through study completion, an average of 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Devarati Mitra, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org